CLINICAL TRIAL: NCT04421755
Title: The Produce Drop: Using Food as Medicine to Lower A1C Levels and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10360
Record Dates: First submitted 2020-04-21; First posted 2020-06-09 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; Hypertension; Nutrition Poor
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Malnutrition

STUDY DESIGN:
Intervention Model Description: A randomized control trial will be used to evaluate the two interventions among a cohort of OU Internal Medicine patients. Clinical and self-report measures will be collected for the intervention arms at four time points: baseline, three months, six months, and nine months and at two time points (baseline and nine months) for the control group. After baseline measures, participants will be randomly assigned to the fruits and vegetables only group, the fruit and vegetables plus cooking classes group, or the control group. This trial will use rolling enrollment, with interventions beginning after the enrollment of enough participants to conduct an effective cooking class. Participants in the intervention groups will receive nine months of free weekly deliveries of fresh fruits and vegetables. Participants in the control group will receive a gift card valued at twenty dollars for each survey completed and an OU gift valued at ten dollars following completion of both surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Produce Only (Experimental): Receives weekly home delivery of fresh fruits and vegetables
  Interventions: Other: Produce delivery
- Produce + Cooking Classes (Experimental): Receives weekly home delivery of fresh fruits and vegetables plus invitation to participate in a series of three small group culinary medicine cooking classes
  Interventions: Other: Produce delivery; Other: Cooking classes
- Control (No Intervention): Control group with no cooking classes or groceries

INTERVENTIONS:
Other: Produce delivery — weekly home delivery of fresh fruits and vegetables
  Arms: Produce + Cooking Classes; Produce Only
Other: Cooking classes — weekly home delivery of fresh fruits and vegetables participants will be invited to participate in a Culinary Medicine cooking series. The OU Culinary Medicine cooking curriculum will involve a 3-part class series designed to build nutrition knowledge and cooking self-efficacy for preparing fresh F/Vs. Each session is ~2 hr. Core nutrition guidelines for blood pressure and blood sugar management will also be emphasized informed by an evidence-based Conceptual Model of Healthy Cooking. Classes will be conducted in small groups (~16 participants) in an established teaching kitchen used by the culinary medicine program. Classes will be facilitated by a professional chef, a healthcare professional (dietitian, medical doctor, or trained medical student), and other support staff, including trained medical, dietetic, and public health students.
  Arms: Produce + Cooking Classes

SUMMARY:
Hypertension and diabetes, which are increasing in prevalence, contribute to significant morbidity and mortality in the U.S. Self-management of these diseases, including adherence to dietary guidelines such as daily fruit and vegetable intake, can improve outcomes, but low-income patients encounter many barriers to adherence, such as food insecurity and poor nutrition literacy. Few clinicians screen for food insecurity, and even when screening is performed, there are few tested clinical response models. This study will evaluate the benefits of fresh fruit and vegetable home delivery program, without and with small-group culinary medicine cooking classes, on blood pressure and glucose control among patients accessing care at the University of Oklahoma Internal Medicine Clinic in Tulsa, OK. The Produce Drop pilot study will evaluate the feasibility and potential health benefits of a clinic-community partnership between OU Internal Medicine and a fresh produce home-delivery service provider, to promote adherence to F/V dietary guidelines among patients with suboptimal blood pressure and blood glucose control. Among half of those assigned to receive food assistance, we will evaluate the additional benefits of participation in 3-session, small-group, hands-on culinary medicine curriculum.

DETAILED DESCRIPTION:
a diet rich in fruits and vegetables, is an essential requirement for optimal blood pressure and glucose control. Clinical practice guidelines for hypertension and diabetes both assign the highest grade of evidence for healthy eating behavior to treat these conditions. Unfortunately, fewer than one-quarter of patients adhere to dietary recommendations, with the largest disparities among lower socioeconomic groups and racial minorities. Patient adherence to nutrition guidelines are deeply hindered by poor access to fresh produce and inadequate knowledge about preparing medically-indicated foods. The proposed Produce Drop pilot study will evaluate the feasibility and potential health benefits of a fresh fruit and vegetable home-delivery program, with and without additional small-group culinary medicine cooking classes, among low-income, Medicaid patients with suboptimal blood pressure and glucose control. Patients (n=100) from OU-Tulsa Schusterman Internal Medicine Clinic will be randomized to 1) a fresh fruit and vegetable home-delivery program, or 2) the same home delivery program with supplementary small-group culinary medicine cooking classes. In addition, we will include a third arm of control patients (n=50) who will receive the standard of care. We will track blood pressure and glucose control in all three groups to determine the comparative impact of each intervention. The proposed pilot study, informed by the Institute for Healthcare Improvement's "Triple Aim" framework, will provide the formative information needed to develop a larger-scale intervention to enhance the patient care experience, improve population health status, and reduce the per capita cost of care.

ELIGIBILITY:
Inclusion:

* English-speaking;
* Between 18 - 64 years old;
* Enrolled in Medicaid at baseline
* Elevated blood pressure and/or A1C scores in the past three months
* Access to regular medical care
* Permission from physician to participate
* Physical home address that can accept grocery deliveries
* Lives inside the grocery service delivery area with no intention to move outside of the service areas in the next 9 months

Exclusion:

* Non-English speaking
* Less than 18 years of age or over 64 years of age
* Serious or terminal illness
* Pregnant or planning to become pregnant in the next 9 months
* Advanced end stage renal disease
* Current enrollment in any other research studies on high blood pressure or diabetes
* No other household member participating in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline, 3 months, 6 months, 9 months
  change scores in systolic blood pressure at each time point
Diastolic blood pressure | Baseline, 3 months, 6 months, 9 months
  change scores in diastolic blood pressure at each time point review include age, medications, insurance, A1c, systolic blood pressure, diastolic blood pressure, weight, height, tobacco use, emergency room use, and hospitalizations. Self-report survey items include demographics, insurance, diabetes/pre-diabetes diagnosis date, hypertension diagnosis date, health literacy, medication adherence and medication scrimping, smoking status (Adult Tobacco Survey), food security (USDA 6-item food security survey), grocery shopping; food access (NEMS-P), consumption of fruit and vegetables from weekly delivery , fruit and vegetable intake (f/v checklist), food preparation/eating at home/eating out behaviors, nutrition-related quality of life (NQOL), cooking knowledge, and cooking confidence.
A1c | Baseline, 3 months, 6 months, 9 months
  change scores in A1C at each time point
Food security | Baseline, 3 months, 6 months, 9 months
  change scores on a food security scale
Food environment | Baseline, 9 months
  change scores on a food environment scale
Fruit and vegetable consumption | Baseline, 9 months
  change scores on a fruit and vegetable consumption scale
Nutrition knowledge | Baseline, 9 months
  change scores on a fruit and vegetable consumption scale
Cooking skills | Baseline, 9 months
  change scores on cooking skills scale

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Wetherill, PhD, Principal Investigator — University of Oklahoma; Brent Beasley, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Schusterman Clinic at the University of Oklahoma Health Science Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No